CLINICAL TRIAL: NCT02171234
Title: A Double-blind, Randomised, Placebo-controlled, Rising Multiple Dose Study to Investigate the Safety, Tolerability, Steady State Pharmacokinetic Profile and CNS Effects of BIA 2-093, in Young Healthy Male Volunteers.
Brief Title: A Double-blind, Randomised, Placebo-controlled, Rising Multiple Dose Study to Investigate the Safety, Tolerability, Steady State Pharmacokinetic Profile and CNS Effects of BIA 2-093
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIA-2093-102
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Results first posted 2015-01-07 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2014-12

CONDITIONS: Epilepsy
Keywords: Epilepsy; BIA 2-093; Eslicarbazepine acetate
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1- 200 mg b.i.d. (twice daily) (Experimental): BIA 2-093 200mg with 200 ml potable water. Identical placebo administered as oral tablets.
  Interventions: Drug: Placebo; Drug: BIA 2-093
- Group 2 - 400 mg b.i.d. (Experimental): BIA 2-093 200mg with 200 ml potable water. Identical placebo administered as oral tablets.
  Interventions: Drug: Placebo; Drug: BIA 2-093
- Group 3- 800 mg o.d. (once daily) (Experimental): BIA 2-093 200mg with 200 ml potable water. Identical placebo administered as oral tablets.
  Interventions: Drug: Placebo; Drug: BIA 2-093
- Group 4 - either 800 mg b.i.d or 1200 mg o.d. (Experimental): BIA 2-093 200mg with 200 ml potable water. Identical placebo administered as oral tablets.
  Interventions: Drug: Placebo; Drug: BIA 2-093

INTERVENTIONS:
Drug: Placebo
  Other Names: PLC, Placebo
Drug: BIA 2-093
  Other Names: ESL, Eslicarbazepine acetate

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of multiple dose regimens of BIA 2-093 in healthy young male volunteers

DETAILED DESCRIPTION:
Single centre, Phase I, double-blind, randomised, placebo-controlled study investigating 4 multiple rising oral doses of BIA 2-093 in 4 groups of 8 young healthy male subjects. Within each group, 2 subjects were randomised to receive placebo and the remaining 6 subjects to receive BIA 2-093. No subject was a member of more than one group. The dose regimens investigated were: 200 mg b.i.d.(twice daily), 400 mg o.d.(once daily; this was changed from 400 mg b.i.d. in protocol amendment 1, on the basis of interim pharmacokinetic analysis of Group 1 data), 800 mg o.d, and 1200 mg o.d. BIA 2-093/placebo was administered orally once daily on Days 1-8, or twice a day (at 12-hour intervals) on Days 1-7 with a final dose in the morning of Day 8. The multiple dose regimens were to be investigated in ascending order. Progression to each higher dose level was only to occur if the previous dose level was deemed by the investigator and the sponsor to be safe and well tolerated.

ELIGIBILITY:
* Inclusion Criteria:
* Adult males aged 18-45 years, with a body mass index (BMI) of 19-28 kg/m2.
* Subjects who were healthy as determined by pre-study medical history, physical examination, 12-lead ECG and EEG.
* Subjects who had clinical laboratory tests acceptable to the investigator.
* Subjects who were negative for HbsAg, anti-HCV and HIV I and II tests at screening.
* Subjects who were negative for drugs of abuse and alcohol tests at screening and admission.
* Subjects who were non-smokers or previous smokers who had not smoked for at least 6 months.
* Subjects who were able and willing to give written informed consent.
* Exclusion Criteria:
* Subjects who did not conform to the above inclusion criteria.
* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had a clinically relevant family history.
* Subjects who had a history of relevant atopy.
* Subjects who had a history of relevant drug hypersensitivity (carbamazepine and
* related compounds).
* Subjects who had a history of alcoholism.
* Subjects who had a history of drug abuse.
* Subjects who consumed more than 28 units of alcohol a week.
* Subjects who had a significant infection or known inflammatory process on screening and/or admission.
* Subjects who had acute gastrointestinal symptoms at the time of screening and/or admission (e.g. nausea, vomiting, diarrhoea, heartburn).
* Subjects who had an acute infection such as influenza at the time of screening and/or admission.
* Subjects who had used prescription drugs within 4 weeks of first dosing.
* Subjects who had used over the counter medication, excluding routine vitamins but including mega dose vitamin therapy, within one week of dosing.
* Subjects who had used any investigational drug and/or participated in any clinical trial within 3 months of admission to this study.
* Subjects who had donated and/or received any blood or blood products within 3 months prior to screening.
* Subjects who were vegetarians, vegans and/or had medical dietary restrictions.
* Subjects who could not communicate reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.
* Subjects who were unwilling or unable to give written informed consent.
* Subjects who had previously received BIA 2-093.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2001-02; Primary Completion 2001-06 (Actual); Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's Drug Research Unit, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: PLC, Placebo
- Group 1 - 200 mg b.i.d.: BIA 2-093 200mg (twice daily)
- Group 2 - 400 mg o.d.: BIA 2-093, ESL, Eslicarbazepine 400mg
- Group 3 - 800 mg o.d.: BIA 2-093, ESL, Eslicarbazepine 800mg
- Group 4 - 1200 mg o.d.: BIA 2-093, ESL, Eslicarbazepine 1200mg
Period: Overall Study
Arm/Group | Placebo | Group 1 - 200 mg b.i.d. | Group 2 - 400 mg o.d. | Group 3 - 800 mg o.d. | Group 4 - 1200 mg o.d.
Started | 8 | 6 | 6 | 6 | 6
Completed | 8 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1 - BIA 2-093 200 mg b.i.d.: BIA 2-093, ESL, Eslicarbazepine acetate 200mg (twice daily)
- Group 2 - BIA 2-093 400 mg o.d.: BIA 2-093, ESL, Eslicarbazepine acetate 400mg
- Group 3 - BIA 2-093 800 mg o.d.: BIA 2-093, ESL, Eslicarbazepine acetate 800mg
- Group 4 - BIA 2-093 1200 mg o.d.: BIA 2-093, ESL, Eslicarbazepine acetate 1200mg
- Total: Total of all reporting groups
Arm/Group | Placebo | Group 1 - BIA 2-093 200 mg b.i.d. | Group 2 - BIA 2-093 400 mg o.d. | Group 3 - BIA 2-093 800 mg o.d. | Group 4 - BIA 2-093 1200 mg o.d. | Total
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 6 | 6 | 6 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 8 | 6 | 6 | 6 | 6 | 32

OUTCOME MEASURES:

1. Secondary Outcome: Cmax
Description: Cmax - Maximum observed plasma concentration
Time Frame: Day 1 and Day 8
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Group 1 - BIA 2-093 200 mg b.i.d. | Group 2 - BIA 2-093 400 mg o.d. | Group 3 - BIA 2-093 800 mg o.d. | Group 4 - BIA 2-093 1200 mg o.d.
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/ml
  Cmax Day 1 | 3086 (1342) | 7827 (1313) | 11074 (1919) | 16071 (2238)
  Cmax Day 8 | 6683 (1576) | 8824 (1411) | 18675 (2613) | 25457 (2746)

2. Secondary Outcome: AUC0-τ
Description: AUC0-τ - Area under the plasma concentration time curve to last measurable time point
  Day 1 - pre-dose, 30, 60, 90, 120, 180 minutes, 4, 6, 7, 8, 12, hours post final dose Day 8 - pre-dose, 30, 60, 90, 120, 180 minutes, 4, 6, 7, 8, 12, 24, 36, 48 and 72 hours post final dose
Time Frame: Day 1 - pre-dose, 30, 60, 90, 120, 180 minutes, 4, 6, 7, 8, 12, hours post final dose Day 8 - pre-dose, 30, 60, 90, 120, 180 minutes, 4, 6, 7, 8, 12, 24, 36, 48 and 72 hours post final dose
Measure: Mean (Standard Deviation); unit: ng.h/ml
Arm/Group | Group 1 - BIA 2-093 200 mg b.i.d. | Group 2 - BIA 2-093 400 mg o.d. | Group 3 - BIA 2-093 800 mg o.d. | Group 4 - BIA 2-093 1200 mg o.d.
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng.h/ml
  AUC0-τ Day 1 | 22163 (6216) | 96262 (17064) | 159492 (21695) | 250426 (27356)
  AUC0-τ Day 8 | 63140 (7997) | 126308 (14833) | 268384 (27683) | 423003 (45952)

3. Primary Outcome: Total Number of Adverse Events
Description: Total Number of Adverse Events.
Time Frame: up to 20 weeks
Measure: Number; unit: Total Number of AE
Arm/Group | Group 1 - BIA 2-093 200 mg b.i.d. | Group 2 - BIA 2-093 400 mg o.d. | Group 3 - BIA 2-093 800 mg o.d. | Group 4 - BIA 2-093 1200 mg o.d. | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Total Number of AE
  All Adverse Events | 9 | 15 | 5 | 12 | 14
  AE Considered Not Related to Treatment | 3 | 2 | 0 | 0 | 1
  AE Considered Possibly Related to Treatment | 6 | 13 | 5 | 12 | 13
  Adverse Events of Mild Severity | 9 | 15 | 4 | 12 | 14
  Adverse Events of Moderate Severity | 0 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Group 1 - BIA 2-093 200 mg b.i.d. | Group 2 - BIA 2-093 400 mg o.d. | Group 3 - BIA 2-093 800 mg o.d. | Group 4 - BIA 2-093 1200 mg o.d.
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/8 | 4/6 | 4/6 | 3/6 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | Group 1 - BIA 2-093 200 mg b.i.d. (N=6) | Group 2 - BIA 2-093 400 mg o.d. (N=6) | Group 3 - BIA 2-093 800 mg o.d. (N=6) | Group 4 - BIA 2-093 1200 mg o.d. (N=6)
Flushing (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Mouth dry (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 1 | 1 | 3
Headache (Nervous system disorders) | 1 | 2 | 1 | 1 | 2
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0
Mucositis NOS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Hepatic enzymes increased (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Skeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Concentration impaired (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Dreaming abnormal (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Somnolence (Psychiatric disorders) | 2 | 0 | 2 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Herpes simplex (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1
Upper resp tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin dry (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other